CLINICAL TRIAL: NCT06939413
Title: Establishing a Sustainable Diabetes Care Management Program Using Continuous Glucose Monitors and Remote Patient Monitoring for Underserved Populations in Safety Net Clinics
Brief Title: Diabetes Management Using Continuous Glucose Monitors and Remote Patient Monitoring in Underserved Populations
Acronym: DCMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Solutions International (Other)
Collaborators: DexCom, Inc. (Industry); Tidepool (Unknown); MAVEN Project (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIS-2024-172
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Uncontrolled type 2 diabetes mellitus; CGM; Remote patient monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Single-arm prospective 24-week study with an optional 28 week extension Patients from a clinic site not involved in the study will be used as case matched controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Other): The participants will be in the intervention arm for 24 weeks with an optional 28 week extension . The intervention being studied is continuous glucose monitoring (CGM) and remote patient monitoring that is being provided as an adjunct to usual diabetes care
  Interventions: Device: Continuous glucose monitor (CGM)

INTERVENTIONS:
Device: Continuous glucose monitor (CGM) — The glucose data from the CGM will help participants to understand the effect of lifestyle and medications on their glucose levels. The glucose levels from the CGM will be remotely monitored. Outreach will be made to participants not reaching glycemic goals. Appropriate adjustments in treatment regimen will be made based on the glucose data obtained from CGM and RPM

SUMMARY:
The goal of this 52 week prospective study is to learn whether a Diabetes Care Management Program using a continuous glucose monitor (CGM) and remotely monitoring (RPM) glucose readings can help improve glucose levels and diabetes related distress in individuals with uncontrolled type 2 diabetes. The CGM and RPM are used as an adjunct to usual care.

The main questions it aims to answer are:

Does use of CGM & RPM improve A1c? Does use of CGM & RPM improve the percent of time spent with glucose levels between 70-180 mg/dl? Does the diabetes care management program improve diabetes related distress?

Participants enrolled in the study will be wearing a CGM. Participants will be able to see the glucose readings from the CGM and see how their glucose level responds to food, physical activity, medications and daily life.

The diabetes primary care team will be remotely monitoring the participant's glucose data from the CGM. They will reach out to the participant to make adjustments in treatment regimen as needed.

Participants will answer a "Problem Areas in Diabetes"questionnaire that asks questions about diabetes related distress.

DETAILED DESCRIPTION:
BACKGROUND & RATIONALE:

Medical Alumni Volunteer Expert Network (MAVEN) Project is a nonprofit organization dedicated to addressing social, racial, and economic inequities in the healthcare system through the power of telemedicine. The project recruits an experienced corps of volunteer medical specialists and connects them virtually with primary care providers (PCPs) at community health centers using a digital health platform. The services provided include medical consults, eConsults, mentoring, and Continuing Medical Education (CME) programs.

Patients with diabetes seen in safety net clinics are more complex with a higher incidence of diabetes related complications and other chronic conditions. PCPs are often overwhelmed and frustrated with managing diabetes in these patients, especially with the lack of glucose data. Continuous glucose monitor (CGM) use provides a complete glucose picture leading to appropriate adjustment in treatment regimen. In addition, individuals wearing a CGM are more likely to modify their physical activity and eating habits based on the real time glucose levels from the CGM.

MAVEN Project has been instrumental in enhancing diabetes management and improving patient outcomes in these safety net clinics, where 1 in 3 persons live in poverty and 63% identify as a racial/ethnic minority.

Given our early success, it became quite apparent that there was an opportunity to develop an evidence-based diabetes care management program incorporating CGM and remote patient monitoring (RPM) that would improve diabetes outcomes in the underserved population with a potential for implementation in other safety net clinics across the country. PCPs at front line clinics have access to endocrinology expertise through MAVEN Project. Remote patient monitoring of CGM data is now possible as over 98% of the FQHCs offer telehealth services as compared to 48 % in 2018.

PRIMARY OBJECTIVE:

To determine if a sustainable diabetes care management program incorporating CGM and RPM can improve glucose levels and diabetes related distress in individuals with diabetes seen at safety net clinics.

SECONDARY OBJECTIVE:

To determine if a sustainable diabetes care management program incorporating CGM and RPM can improve clinician and patient satisfaction.

STUDY DESIGN:

This is a single-arm prospective 24-week study with an optional 28 week extension designed to investigate the effect of a sustainable diabetes care management program incorporating CGM and RPM on improving glucose levels, diabetes related distress and patient satisfaction in individuals with diabetes seen at safety net clinics. PCP satisfaction will also be assessed. Patients from a clinic site not involved in the study will be used as case matched controls.

All eligible subjects will start on CGM & RPM. Participants will use "guided experiments "during the first 7 to 10 days to understand the effects of food and physical activity on their glucose levels., Participants will follow up with the diabetes primary care team in 10-14 days to review the glucose data.

It is anticipated that about 20% of participants will require insulin and 80% will be on non-insulin treatment. Participants on insulin will continue real time CGM wear throughout the 52-week study. Participants not on insulin will wear real time CGM for the first 12 weeks and intermittently thereafter. All participants will be educated on the use of CGM to help manage their diabetes.

The RPM dashboard will be reviewed weekly, and outreach made to participants with low time in range 70-180 mg/dl (TIR) or no sensor data. CGM and RPM data will be used to adjust the treatment regimen.

CME will be provided by MAVEN Project on topics that are crucial for the PCPs to effectively manage diabetes. A PCP baseline educational needs assessment will be obtained to help guide the timing and necessity of the various CME sessions. Educational sessions will be provided for ancillary staff.

Endocrinology expertise will be provided through e-consults to MAVEN endocrinologists for specific patient management questions. MAVEN Endocrinologists will provide additional support through biweekly meetings with the clinic diabetes champion and monthly study site meetings.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older with Type 2 diabetes AND
* A1c > 8%

Exclusion Criteria:

* Pregnancy (participant-reported)
* Previous real time CGM use for more than 6 weeks in the last 3 months
* Use of steroids
* Active cancer treatment
* Terminal illness
* Dementia, mental impairment
* Type 1 diabetes
* End stage renal disease, on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in A1c | Baseline, 12, 24, 36 and 52 weeks
  A1c is a blood test that measures the average glucose level over the previous 2 to 3 months. A normal A1c is 5.7 to 6.4%. The usual goal for most people with diabetes is < 7% or as close to normal as possible without low glucose levels
Change in time in range (TIR) | Baseline, 6, 12, 24, 36 and 52 weeks
  TIR measures the percentage of glucose values between 70-180 mg/dl ie the percentage of time spent between 70-180 mg/dl . The usual goal for most individuals with diabetes is to have TIR > 70%
Change in Problem Areas in Diabetes (PAID) score | Baseline, 12, 24 and 52 weeks
  PAID is a 20 point questionnaire that assesses diabetes related distress. A lower score indicates less diabetes related distress. A score of > 40 indicates significant diabetes related distress. Typically the PAID score decreases in response to diabetes care management. An extremely low score (0-10) combined with high glucose levels may be indicative of denial. The score can range from 0 to 125.

SECONDARY OUTCOMES:
Change in time above range (TAR) | Assessed at baseline, 6, 12, 24, 36 and 52 weeks
  TAR measure the percent of time with glucose levels > 180 mg/dl. The usual goal for diabetes is < 25%
Change in time below range (TBR) | Assessed at baseline, 6, 12, 24, 36 and 52 weeks
  TBR measure the percent of time with glucose levels < 70 mg/dl. The usual goal for diabetes is < 4%
Change in Glucose Management Indicator (GMI) | Assessed at baseline, 6, 12, 24, 36 and 52 weeks
  GMI provides an estimate of the A1c level based on the average glucose levels measured by a continuous glucose monitor (CGM) over the previous 14 days A normal GMI is 5.7 to 6.4% . The usual goal for diabetes is < 7% or as close to normal as possible without a low glucose
Patient Satisfaction Survey | Assessed at 12, 24 and 52 weeks
  This is a survey that measures the patient's satisfaction with the diabetes care management program. The questions use a 5-point Likert scale with a higher score indicating satisfaction with the program . The score can range from 7 to 35.
Change in Primary care provider (PCP) Satisfaction | Assessed at baseline , 24 and 52 weeks
  The survey assesses the PCP satisfaction with how diabetes care is delivered in the clinic. The questions use a 5-point Likert scale with the score ranging from 5 to 15. A higher score indicates satisfaction with the program.

CONTACTS AND LOCATIONS:
Overall Officials: Sushma Reddy, MD, Principal Investigator — Diabetes Solutions International
Locations (1):
- Community Health Center of Franklin County, Greenfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-01-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT06939413/ICF_000.pdf